CLINICAL TRIAL: NCT00719537
Title: Oral Progesterone and Low Dose Aspirin in the Prevention of Preeclampsia in Patients With a Prior History of Preeclampsia: A Prospective, Randomized Clinical Trial
Brief Title: Oral Progesterone and Low Dose Aspirin in the Prevention of Preeclampsia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to find qualifying participants
Sponsor: John Uckele (Other)
Responsible Party: Sponsor-Investigator, John Uckele, Medical Doctor, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-054
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Preeclampsia
Keywords: preeclampsia; progesterone; aspirin; prevent; soluble fms-like tyrosine kinase (sFlt-1); Placental Growth Factor (PlGF); risk
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin plus Placebo Oral Tablet (Placebo Comparator): Drug: Aspirin 81 mg, given orally once per day Drug: Placebo tablet given orally, once a day
  Interventions: Drug: Aspirin; Drug: Placebo Oral Tablet
- Aspirin plus Progesterone (Active Comparator): Drug: Aspirin 81mg, given orally once per day Drug: Progesterone 200mg given orally, once a day
  Interventions: Drug: Aspirin; Drug: Progesterone

INTERVENTIONS:
Drug: Aspirin — Aspirin 81 mg once a day
Drug: Placebo Oral Tablet — Placebo 1 tab Daily
  Arms: Aspirin plus Placebo Oral Tablet
Drug: Progesterone — Oral Progesterone 200 mg Twice Daily
  Arms: Aspirin plus Progesterone

SUMMARY:
This study investigates whether low dose aspirin combined with progesterone will decrease the risk of preeclampsia in pregnant women with a history of preeclampsia in a previous pregnancy.

DETAILED DESCRIPTION:
Recent advances have shown that certain proteins may be present in a pregnant woman's blood very early in pregnancy which can predict who is at the highest risk for developing preeclampsia. These proteins can be measured and may be used to predict a woman's risk of developing preeclampsia.

Special placental cells called endovascular cytotrophoblasts are needed in the early formation of the placenta. These placental cells invade the maternal blood vessels in the formation of the maternal-placental blood interface. Human Leukocytes Antigen-G (HLA-G) is a protein produced by the placental cells and prevents these special cells from being rejected by the mother's immune system. Recent studies have indicated that the level of HLA-G is decreased in placentas from mothers with preeclampsia. Progesterone, a naturally occurring hormone produced in pregnancy, has been shown to increase the production of HLA-G in the placental cytotrophoblast cells.

In regards to the treatment of preeclampsia, studies have shown that low dose aspirin if given to mothers who have had severe early preeclampsia, lowers the risk for having preeclampsia again. This study aims to show that low dose aspirin combined with progesterone will decrease the risk of preeclampsia in pregnant women with a history of preeclampsia in a previous pregnancy. Data generated will determine levels and ratios of blood proteins that are predictive of preeclampsia at specific gestational ages.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients with a previous history of preeclampsia in the immediate preceding pregnancy.
* 18 to 45 years of age will be included.

Exclusion Criteria:

* Patients with chronic hypertension
* children (age < 17 years)
* Patients that are currently taking anti-psychotics or Selective Serotonin Re-uptake Inhibitors
* patients on medications which may be detrimental to the study interpretation will also be excluded at the principal investigator's discretion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Uckele, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No study data is available, will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin and Placebo: Aspirin and placebo: Aspirin 81mg once daily and placebo once daily
- Aspirin and Progesterone: aspirin 81 mg once a day oral progesterone 200mg twice daily
Period: Overall Study
Arm/Group | Aspirin and Placebo | Aspirin and Progesterone
Started | 2 | 1
Completed | 1 | 0
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin and Placebo | Aspirin and Progesterone | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants] — 18-50 years, female
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 1 | 3
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Preeclampsia
Description: Number of Participants with preeclampsia in second and third trimester of pregnancy.
Time Frame: second and third trimester of pregnancy
Population: 1 Participant withdrawn in aspirin and placebo group, one participant lost to followup in aspirin and progesterone group.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin and Placebo | Aspirin and Progesterone
Number analyzed (Participants) | 1 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Aspirin and Placebo: Aspirin and placebo: Aspirin 81mg once daily and placebo
- Aspirin and Progesterone: Aspirin and progesterone: aspirin 81 mg once a day oral progesterone 200mg twice daily
Arm/Group | Aspirin and Placebo | Aspirin and Progesterone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No